CLINICAL TRIAL: NCT01525095
Title: Detecting Infections Rapidly and Easily for Candidemia Trial (DIRECT)-Part 1 (Prospective Collection and Freezing of Whole Blood Specimens)
Brief Title: Detecting Infections Rapidly and Easily for Candidemia Trial (DIRECT)
Acronym: DIRECT
Status: Completed | Type: Observational
Sponsor: T2 Biosystems (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00030
Record Dates: First submitted 2012-01-25; First posted 2012-02-02 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Candidemia
Keywords: Candida; Diagnostic Assay; Blood culture; Sepsis; T2 Magnetic Relaxation
MeSH Terms: conditions — Candidemia; Torulopsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood specimens, in addition to bacterial and fungal species isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Candida Positive Patients: Symptomatic adult patients, confirmed via concordant diagnostic blood culture and species identification and subsequent second blood culture results and species identification that are Candida positive
- Candida Negative Patients: Hospitalized adult patients, confirmed via concordant diagnostic blood culture with subsequent species identification and subsequent second blood culture with subsequent species identification that are Candida negative

SUMMARY:
The purpose of this study is to assure the uniform collection, handling, storage and transport of patient whole blood specimens and associated information to support validation of the T2 Candida Assay.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's authorized representative must be able to understand, read and sign the study specific informed consent form after the nature of the study has been fully explained to them.
2. For Group A,

   * Males and females 18 - 95 years of age.
   * Subject is confirmed to have fungemia as evidenced by a positive diagnostic blood culture and subsequent species identification.
3. For Group B,

   * Males and females 18 - 95 years of age.
   * Subject is hospitalized with a medical problem other than fungemia, or is being treated as an outpatient for some non-infection-related condition, and
   * Subject is confirmed to not have fungemia as evidenced by diagnostic blood culture and subsequent species identification.

Exclusion Criteria:

1. Use of any novel (i.e. not commercially available) drug compound within 30 days prior to the collection of T2 blood specimens.
2. Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have undergone a diagnostic blood culture.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Candida Positive patients | 3-5 days post blood culture
  Number of Candida Positive patients based on concordant, sequential blood culture results and a positive T2 signal

SECONDARY OUTCOMES:
Number of Candida Negative Patients | 3-5 days post blood culture
  Number of Candida Negative patients based on concordant, sequential blood culture results and a negative T2 signal

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pappas, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - University of Houston College of Pharmacy, Houston, Texas

REFERENCES:
- [Derived] Clancy CJ, Pappas PG, Vazquez J, Judson MA, Kontoyiannis DP, Thompson GR 3rd, Garey KW, Reboli A, Greenberg RN, Apewokin S, Lyon GM 3rd, Ostrosky-Zeichner L, Wu AHB, Tobin E, Nguyen MH, Caliendo AM. Detecting Infections Rapidly and Easily for Candidemia Trial, Part 2 (DIRECT2): A Prospective, Multicenter Study of the T2Candida Panel. Clin Infect Dis. 2018 May 17;66(11):1678-1686. doi: 10.1093/cid/cix1095. PMID 29438475
- [Derived] Clancy CJ, Nguyen MH. Finding the "missing 50%" of invasive candidiasis: how nonculture diagnostics will improve understanding of disease spectrum and transform patient care. Clin Infect Dis. 2013 May;56(9):1284-92. doi: 10.1093/cid/cit006. Epub 2013 Jan 11. PMID 23315320